CLINICAL TRIAL: NCT01179750
Title: The Use of Ultrasonic Coagulating Shears Compared to Monopolar Electrocautery in Open Gastric Cancer Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Jae Moon Bae, Samsung Medical Center, Sungkyunkwan University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-08-089
Record Dates: First submitted 2010-07-27; First posted 2010-08-11 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Stomach Cancer; Gastrectomy; Ultrasonic Coagulating Shears
Keywords: Ultrasonic coagulating shears in gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Ultrasonic Coagulating Shears group (No Intervention): the one arm: operated group without using Ultrasonic coagulation shears during gastrectomy;
- ultrasonic coagulation shears group (Experimental): the other arm: operated group using ultrasonic coagulation shears during gastrectomy
  Interventions: Device: Ultrasonic Coagulating Shears

INTERVENTIONS:
Device: Ultrasonic Coagulating Shears — comparison of operated groups between with Ultrasonic Coagulating Shears and without them.
  Other Names: Harmonic Ace
  Arms: ultrasonic coagulation shears group

SUMMARY:
Ultrasonic coagulating shears are made for performing for cutting and hemostasis at once during operation. It was proved that a laparoscopic gastric resection showed significantly shorter operative time and less work load distribution, and more stability of bleeding than before an introduction of ultrasonic coagulating shears .

In an open gastric cancer surgery, ultrasonic coagulating shears have been often used for lymph node dissection or cutting of small vessels in some hospitals in Korea. However its usefulness or effectiveness has not been fully proved. There was only one report about using ultrasonic coagulating shears in open gastrectomy. The report contained small number of subjects and surgical procedures were different from the investigators.

The investigators expect to reduce operative time and blood loss with ultrasonic coagulating shears. Ultrasonic coagulating shears will also enable us to dissect lymph node with closure of lymphatics. This may reduce the amount of drainage fluid from peritoneal cavity and shorten the removal time of a drain, which will also shorten the hospital stay.

The objective of this study is to evaluate the safety and benefit of ultrasonic coagulating shears in open gastrectomy including usefulness and effectiveness by a randomized controlled, prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of gastric cancer
* The patient who agrees to participate in this study by signing the informed consent form

Exclusion Criteria:

* The patient who refuse to participate in this study
* Have simultaneously other cancer
* Underwent cancer therapy at past time
* Have bleeding disorder, coagulation disorder, chronic disease (e.g.heart failure, cardiovascular disease, active hepatitis)
* Have a previous upper gastrointestinal surgery

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-04 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
operation time | 2 weeks later after operation
  operation time: a time from the opening of peritoneal cavity to the retrieval of specimen
amount of blood loss | 2 weeks later after operation
  amount of blood loss: an amount of blood loss during operation time

SECONDARY OUTCOMES:
C-reactive protein | post operative day #0, #1, #5
total lymphocyte count | post operative day #0, #1, #5
postoperative complications | 4 weeks later after operation
drainage from peritoneal cavity during hospital | 2 weeks later after operation
  amount of drainage: an amount of postoperative draining fluid from peritoneal cavity during hsopital

CONTACTS AND LOCATIONS:
Overall Officials: Jae Moon Bae, MD., Ph.D., Principal Investigator — Samsung Medical Center, Sungkyunkwan University
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Tsimoyiannis EC, Jabarin M, Tsimoyiannis JC, Betzios JP, Tsilikatis C, Glantzounis G. Ultrasonically activated shears in extended lymphadenectomy for gastric cancer. World J Surg. 2002 Feb;26(2):158-61. doi: 10.1007/s00268-001-0199-9. Epub 2001 Dec 4. PMID 11865342